CLINICAL TRIAL: NCT02447627
Title: A Study of Methodologies to Measure Blood Flow and Oxygenation as Potential Biomarkers in Adults With Sickle Cell Disease
Brief Title: Study of Methodologies to Measure Blood Flow and Oxygenation in Adults With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: 996SC001
Record Dates: First submitted 2015-04-16; First posted 2015-05-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-08

CONDITIONS: Healthy; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for hematology, blood chemistry, and venous blood gas analysis. Blood samples will also be used for exploratory biomarker development specific to SCD.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part A: Cohort 1- Participants with severe SCD (4-10 VOC/year) Cohort 2- Participants with milder SCD (<4-10 VOC/year) Cohort 3- Healthy volunteers Part A and B can occur in parallel
- Part B: Adults with SCD receiving chronic red blood cell exchange transfusion Part A and B can occur in parallel

SUMMARY:
The purpose of the study is to determine whether imaging techniques, such as magnetic resonance imaging (MRI), near infrared spectroscopy (NIRS), laser speckle contrast imaging (LSCI), and optical imaging (OI), can detect differences in blood flow and oxygen levels in different organ systems of participants with sickle cell disease (SCD). Differences in blood flow and oxygen levels detected by these techniques will be evaluated to determine their utility as biomarkers of clinical disease pathophysiology.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have a diagnosis of SCD confirmed by hemoglobin analysis.
2. Be in stable clinical condition, as determined by the Investigator.

   Subjects enrolled in Part B must also meet the following eligibility criterion at Screening:
3. Receiving scheduled standard of care RBC exchange transfusion therapy, with ≥3 transfusions already received.
4. Be deemed healthy, as determined by the Investigator, based on the physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory measurements.

Key Exclusion Criteria:

1. Inability to lie still for ≥5 minutes, claustrophobia sufficient to interfere with generating reliable MRI scans, body weight exceeding 320.0 lbs., or girth exceeding the magnet bore.
2. Presence of a metal device affected by MRI (e.g., any type of electronic, mechanical or magnetic implant, cardiac pacemaker, aneurysm clips, implanted cardiac defibrillator) or potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) which would be a contraindication for MRI.
3. Acute pain crisis requiring hospitalization, with a discharge ≤4 weeks prior to the first imaging visit, or when determined by the Investigator to not be at steady state.
4. Recent (≤3 months) treatment with hydroxyurea therapy.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with mild to severe VOC
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Blood flow in the brain of adults with severe SCD (4-10 vaso-occlusive crises [VOC]/ year) compared to healthy adults without SCD as assessed by MRI-ASL (arterial spin labeling) | Up to day 18 post screening visit

SECONDARY OUTCOMES:
Kidney blood flow rates as assessed by MRI-SWI (susceptibility-weighted imaging) | Up to day 21 post screening visit
Skeletal muscle blood flow rates as assessed by NIRS | Up to day 21 post screening visit
Skin blood flow rates as assessed by LSCI | Up to day 21 post screening visit
Retinal blood flow rates as assessed by OI | Up to day 21 post screening visit
Total oxygen levels in the brain as assessed by MRI-ASL | Up to day 21 post screening visit
Total oxygen levels in the kidney as assessed by MRI-SWI | Up to day 21 post screening visit
Total oxygen levels in the muscle as assessed by NIRS | Up to day 21 post screening visit
Total oxygen levels in the skin as assessed by LSCI | Up to day 21 post screening visit
Total oxygen levels in the retina as assessed by OI | Up to day 21 post screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (1):
- Research Site, Detroit, Michigan, United States